CLINICAL TRIAL: NCT04709263
Title: Heart Failure Patients Registry A Prospective Observational Multicenter Registry of Patients With Chronic Heart Failure in the Population of the Russian Federation (PRIORITY-HF)
Brief Title: Heart Failure Patients Registry
Acronym: Priority-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00323
Record Dates: First submitted 2020-12-22; First posted 2021-01-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
This study is a multicenter non-interventional observational prospective registry. This non-interventional study (NIS) does not imply any intervention into a routine clinical practice, including choice of treatment modality or special methods of investigation. The study will include only those patients who sign the informed consent form (ICF) after explanation of the study objectives and methods by the study physician.

Planned study population consists of 20 000 adult outpatients with HF. All patients with HF who signed an ICF will be included to this study. Planned number of study sites is 150 outpatient centers in about 50 regions (in order to describe characteristics of outpatients with HF in different regions in the most comprehensive way).

Expected inclusion period duration - 24 months OR reaching 20 000 patients, if this takes less than 24 months. Planned follow-up period duration for 1 patient is about 52 weeks (12 months), which includes 3 visits (visit 1 - inclusion; visit 2 - approximately 6 months after inclusion; visit 3 - approximately 12 months after inclusion)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of inclusion;
2. Signed and dated written informed consent in accordance with ICH GCP and local law prior to inclusion in the study;
3. Documented diagnosis of HF (according to Clinical Guidelines "Chronic Heart Failure", 2020, approved by MoH of RF) with typical symptoms/signs of HF consistent with I-IV functional classes of HF according to NYHA classification.

Exclusion Criteria:

1. The absence of signed ICF;
2. The participation in any randomised controlled trial within 3 months before the inclusion in this study or during the participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional multicenter observational study will include 20,000 adult outpatients with HF who are monitored and treated by cardiologists or internal medicine specialists. In the study, patients will be followed up for about 12 months after being included in approximately 150 clinical centers in Russia. This NIS does not imply any intervention in routine clinical practice, including choice of treatment modality or special methods of investigation. It is planned to include all patients with CHF, who gave their informed consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 19990 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Mean age | Baseline
  At baseline of this study
Proportion of men and women | Baseline
  At baseline of this study
Proportion of patients with negative lifestyle factors | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different etiology of CHF | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with a history of HF comorbidities and conditions of special interest | Baseline
  At baseline of this study
Mean duration of comorbidities listed in previous paragraph (p. 5) (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different chronic comorbidities | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with history of COVID-19 | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with vaccination | Baseline
  At baseline of this study
Proportion of patients with different types of HF based on LVEF | Baseline
  At baseline of this study
Proportion of patients with T2DM comorbid with different types of HF based on LVEF | Baseline
  At baseline of this study
Mean HbA1c (for patients with T2DM) (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF); | Baseline
  At baseline of this study
Proportions of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different levels of HbA1c (for patients with T2DM) | Baseline
  At baseline of this study
Mean BMI (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different BMI levels | Baseline
  The BMI will be calculated using a formula based on the patient's anthropometric data collected at visit q (height measured in meters and body weight measured in kilograms). BMI (kg / m2) is calculated using the formula: BMI = weight (kg) / (height2 (m2))
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different functional classes of CHF according to NYHA classification based on patient symptoms of HF | Baseline
  At baseline of this study
Mean NT-proBNP level (or BNP) | Baseline
  NT-proBNP is measured in pg / mL. At baseline of this study
Mean heart rate (HR) (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF); | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different functional classes of HF according to SHOKS level | Baseline
  1. Functional Class I - ≤3 points;
  2. Functional Class II - from 4 to 6 points;
  3. Functional Class III - from 7 to 9 points;
  4. Functional Class IV - more than 9 points;
  At baseline of this study.
Mean SBP (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  SBP - Systolic blood pressure. At baseline of this study.
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with SBP | Baseline
  1. <90 mm Hg;
  2. 90-99 mm Hg;
  3. 100-109 mm Hg;
  4. 110-119 mm Hg;
  5. 120-139 mm Hg;
  6. 140-159 mm Hg;
  7. ≥160 mm Hg;
  At baseline of this study
Mean Diastolic blood pressure (DBP) (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with DBP | Baseline
  1. <90 mm Hg;
  2. ≥90 mm Hg;
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with concomitant CKD of different stages | Baseline
  eGFR = 141 x min(SCr/κ, 1)^α x max(SCr/κ, 1)^-1.209 x 0.993^Age x 1.018 [if female] x 1.159 [if Black], where eGFR (estimated glomerular filtration rate) = mL/min/1.73 m^2, SCr (standardized serum creatinine) = mg/dL, κ = 0.7 (females) or 0.9 (males), α = -0.329 (females) or -0.411 (males), min = indicates the minimum of SCr/κ or 1, max = indicates the maximum of SCr/κ or 1, age = years.
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with CKD and different levels of albumin-to-creatinine ratio in a spot urine sample | Baseline
  1. <30 mg/g;
  2. 30-300 mg/g;
  3. >300 mg/g;
  At baseline of this study
Proportion of patients (in total sample, in subgroups of patients with HFrEF, HFmEF and HFpEF, in sub-subgroups of patients with CKD and without CKD) with concomitant hyperkalemia (K+ level >5,5 mmol/L) | Baseline
  At baseline of this study
Proportion of patients (in total sample, in subgroups of patients with HFrEF, HFmEF and HFpEF, in sub-subgroups of patients with CKD and without CKD) with concomitant hypokalemia (K+ level <3,5 mmol/L) | Baseline
  At baseline of this study
Mean LVEF (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Mean K+ level (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Mean Na+ level (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Mean hemoglobin level (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different rhythm | Baseline
  1. Sinus rhythm;
  2. AF / AFl;
  3. Pacemaker rhythm;
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with different QRS duration | Baseline
  1. <130 ms;
  2. 130-150 ms;
  3. >150 ms;
  At baseline of this study
Proportion of patients receiving different classes of drugs for treatment of HF | Baseline
  * ACE inhibitors (duration, dosage, proportion of patients receiving: <50% of target dose, 50-100% of target dose, ≥100% of target dose);
  * B-blockers (duration, dosage, proportion of patients receiving: <50% of target dose, 50-100% of target dose, ≥100% of target dose);
  * ARBs (duration, dosage, proportion of patients receiving: <50% of target dose, 50 100% of target dose, ≥100% of target dose);
  * MRAs (duration, dosage, proportion of patients receiving: <50% of target dose, 50 100% of target dose, ≥100% of target dose);
  * ARNI (duration, dosage, proportion of patients receiving: <50% of target dose, 50 100% of target dose, ≥100% of target dose);
  At baseline of this study
Proportion of patients with HFrEF with implantable devices | Baseline
  * Implantable cardioverter-defibrillator (ICD) (recommended; implanted);
  * Cardiac resynchronisation therapy (CRT) (recommended; implanted);
  * CRT with defibrillation (CRT-D) (recommended; implanted);
  * Left ventricular assist device (LVAD);
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with cardiac surgery and endovascular procedures | Baseline
  * Revascularisation with PCI;
  * Revascularisation with CABG;
  * Valvular surgery;
  * Heart transplantation;
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) receiving dual disease-modifying therapy | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) receiving triple disease-modifying therapy | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) receiving quadruple disease-modifying therapy | Baseline
  At baseline of this study
Proportion of patients (in total sample and subgroups of patients with HFrEF, HFmEF and HFpEF) with CHF receiving different classes of glucose lowering drugs and their combinations for T2DM treatment | Baseline
  * Modification of diet and lifestyle only;
  * Metformin;
  * Sulfonylureas;
  * Inhibitors of dipeptidyl peptidase-4 (iDPP4);
  * iSGLT2;
  * Glucagon-like peptide-1 receptor agonists (GLP1 RA);
  * Acarbose;
  * Insulins.
  At baseline of this study

CONTACTS AND LOCATIONS:
Locations (65):
- Russia (65):
  - Research Site, Akhtubinsk, Astrakhan Oblast
  - Research Site, Stary Oskol, Belgorod Oblast
  - Research Site, Gurievsk, Kaliningrad Oblast
  - Research Site, Rodniki Settlement, Kaliningrad Oblast
  - Research Site, Korolyov, Moscow Oblast
  - Research Site, Lyubertsy, Moscow Oblast
  - Research Site, Pushchino, Moscow Oblast
  - Research Site, Bor, Nizhniy Novgorod Region
  - Research Site, Beslan, North Ossetia-Alania
  - Research Site, Zubova Polyana Settlement, Respublika Mordoviya
  - Research Site, Aramil, Sverdlovsk Oblast
  - Research Site, Arkhangelsk
  - Research Site, Astrakhan
  - Research Site, Barnaul
  - Research Site, Bataysk
  - Research Site, Belgorod
  - Research Site, Bryansk
  - Research Site, Cheboksary
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Kirov
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Kursk
  - Research Site, Lipetsk
  - Research Site, Makhachkala
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Oryol
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Stavropol
  - Research Site, Surgut
  - Research Site, Syktyvkar
  - Research Site, Tambov
  - Research Site, Tula
  - Research Site, Tver'
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Ulyanovsk
  - Research Site, Vladimir
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
  - Research Site, Yoshkar-Ola

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00323&attachmentIdentifier=b0416c6d-623f-4b5e-9e24-0380c2cb9fb4&fileName=Redacted_CSR_Synopsis_D184R00323.pdf&versionIdentifier=